CLINICAL TRIAL: NCT06517238
Title: Development and Evaluation of a New Digital Communication Tool Between Dentists and Orthodontists to Improve Oral Prevention for Patients With Multi-bracket Treatment
Brief Title: A New Digital Communication Tool Between Dentist and Orthodontist to Improve Dental Prevention
Acronym: ComDentODFPrev
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2023Ao001
Record Dates: First submitted 2023-12-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-04

CONDITIONS: Reduction in DMFT Index and Plaque Index in Patients at the Treatment Completion, an Average of 4 Years; DMFT Index, ICDAS Score, Dental Plaque Index, Communication, Prevention, Dentist, Orthodontist
Keywords: Carious lesions; individual caries-risk; plaque index; prevention; communication; dentist; orthodontist; ICDAS
MeSH Terms: conditions — Communication; Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Children starting a multi-brackets orthodontic treatment in the oral medicine department of University Hospital of Reims from January 2024. These childrens benefit from semi-annual appointment to analyze their oral health and their individual caries-risk by dentist. Moreover, these results will be communicated with a digital tool to orthodontist who can choose to adapt the orthodontic treatment of these childrens.
  Interventions: Other: There is no intervention
- Control group
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — Observal Study.There is no intervention

SUMMARY:
Dentists and orthodontists of the oral medicine department of Reims University Hospital noted that many children presented white spots around orthodontic brackets, or decays at the end of their multi-brackets orthodontic treatment. These defects required dental cares and sometimes led to dental avulsions. These situations highlighted a poor oral hygiene of children (poorly done or insufficient dental brushing), a lack of oral prevention of their dentist and/or orthodontist, or even a lack of communication between these two practitioners.

The objective of this study is to evaluate if a regular prevention and a specific communication between dentist and orthodontists could reduce the individual caries-risk of patients with multi-brackets orthodontic treatment. During all the orthodontic treatment, a semi-annual oral prevention consultation will be established for each patient, and a digital communication tool will be made available to dentists and orthodontists to facilitate their exchanges.

The study population consists of children under 18 years-old when laying multi-brackets orthodontic treatment.

The study population consists of children aged 8 to 18 years-old (at the start of treatment) treated with multi-brackets orthodontic treatment. The study population is divided in two groups: (i) a control group corresponding to children not benefiting from regular oral preventive follow up monitoring and completing their orthodontic treatment during the year in 2024; (ii) a study group composed of children starting their orthodontic treatment during the year in 2024 and benefiting from regular oral prevention every 6 months, up to four years.

Several parameters will be evaluated from patient medical records: the caries index, the ICDAS score, the plaque index, the oral hygiene and food habits. Concerning the study group, a new digital communication tool will be made available to the dentist and the orthodontist to monitor the oral hygiene of patients. An evaluation of the oral hygiene will be done every 6 months.

The expected outcomes of this study concern the interest of (i) a bi-annual prevention consultation to reduce caries risk, (ii) a regular communication between practitioners to adjust the orthodontic treatment according to the individual caries-risk.

The expected hypothesis is to decrease the patient's caries and plaque indexes in the study group.

DETAILED DESCRIPTION:
The study population consists of children under 18 years-old when laying multi-brackets orthodontic treatment in the oral medicine department of Reims University Hospital. This population is distributed into 2 groups. The control group consists in children having completed their orthodontic treatment by December 2024, (n=30). The study group consists in children starting their orthodontic treatment during 2024 and benefiting from semi-annual oral prevention during four years-treatment. Moreover, their dentists and orthodontists will be able to access a digital communication tool to facilitate their exchanges. The number of patients in the study group will depend on the number of the patients in the control group.

The study protocol was approved by a regulatory agreement of the RGPD (register of processing activities) of Reims University Hospital since 14/11/23. All data will be anonymized. These data correspond to those that are systematically and usually collected by professionals during the orthodontic treatment. They will be stored in a secure computer located in the oral medicine department. The aim of the study and clinical procedures will be explained to the parents and the children to obtain their informed consent.

Data collected for control group at the treatment completion, an average of 4 years: put out the treatment:

* Sex: Girl/Boy/Non-Registered
* Date of birth (month/year) / age
* Processing end date
* Regular orthodontic appointment
* Socio-Professional Category (PCS 2020 level 1 nomenclature: 6 levels INSEE) : farmers; artisans, traders and business leaders; executives and higher intellectual professions; intermediate professions ; employees ; workers
* Decayed, missing and filled teeth index (DMFT Index)
* ICDAS score (International Caries Detection and Assessment System)
* Decays under dental restauration
* Modified orthodontic plaque index (MOP Index)
* Individual carious risk (based on HAS-France):

  * Regular brushing
  * Manual or electric brushing
  * Presence of snacking and soda
  * Taking long-term sweet or medication causing hyposialia
  * Presence of dental plaque visualized by dental plaque disclosing tablet
  * Presence of dental plaque visible without dental plaque disclosing tablet
  * Presence of enamel demineralization
  * Presence of caries lesions (dentin involvement) and/or reversible initial lesions (enamel involvement)
  * Serrated grooves in molars
  * Grooves treated by Sealent
  * Fluoride varnish
* Presence of gingival hyperplasia

Data collected for study group during each consultation before the orthodontic treatment and followed every 6 months, up to 4 years:

* Appointment date
* Sex: Girl/Boy/Non-Registered
* Date of birth (month/year) / age
* Regular follow-up with a dentist
* Socio-Professional Category (PCS 2020 level 1 nomenclature: 6 levels INSEE) : farmers; artisans, traders and business leaders; executives and higher intellectual professions; intermediate professions ; employees ; workers
* Decayed, missing and filled teeth index (DMFT Index)
* ICDAS score (International Caries Detection and Assessment System)
* Plaque Index Silness et Loe before treatment
* Modified orthodontic plaque index (MOP Index) as soon as the treatment is applied
* Molar Incisor Hypomineralization (MIH): degree of severity (moderate - severe), type of teeth affected (molars - incisors), number of teeth treated
* Amelar abnormality: incisal dysplasia, number of teeth treated
* Individual carious risk (based on HAS-France):

  * Regular brushing
  * Manual or electric brushing
  * Presence of snacking and soda
  * Taking long-term sweet or medication causing hyposialia
  * Presence of dental plaque visualized by dental plaque disclosing tablet
  * Presence of dental plaque visible without dental plaque disclosing tablet
  * Presence of enamel demineralization
  * Presence of caries lesions (dentin involvement) and/or reversible initial lesions (enamel involvement)
  * Serrated grooves in molars
  * Grooves treated by Sealent
  * Fluoride varnish
* Presence of gingival hyperplasia
* Need for prevention and/or care sessions

ELIGIBILITY:
Inclusion criteria:

Patients aged under 18 years old when laying treatment. They required multi-brackets orthodontic treatment in the oral medicine department of the Reims University Hospital

Exclusion criteria:

* children under 8 years old
* Patients requiring other orthodontic treatment than multi-brackets,
* Patients requiring any orthodontic treatment
* disabled (with a loss of autonomy that don't allow proper brushing)
* dental pathologies like amelogenesis imperfect, dentinogenesis imperfect, ectodermal dysplasia.

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients were 8 and 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure of DMFT index | every 6 months, up to 4 years
  Number of Decayed, Missing due to caries, and Filled Teeth
Measure of plaque index (Silness and Loe) | every 6 months, up to 4 years
  * Score 0 : absence of microbial plaque
  * Score 1 : film of bacterial plaque invisible to the naked eye; but thin film of microbial plaque along the free gingival margin collected with a probe
  * Score 2 : moderate accumulation with plaque in the sulcus visible to naked eye
  * Score 3 : large amount of plaque visible in sulcus or pocket along the free gingiva margin up to 2mm thick.
Modified Orthodontic Plaque index (MOP) | every 6 months, up to 4 years
  * Score 0 : no plaque.
  * Score 1 : accumulation of mesial and/or distal plaque at the base of the attachment.
  * Score 2 : accumulation of mesial, distal, incisal and/or cervical plaque at the base of the attachment.
  * Score 3 : continuous plaque accumulation from the marginal gingiva to the base of the attachment.
  * Score 4 : complete coverage by the plaque.
Measure of ICDAS score | every 6 months, up to 4 years
  * 0 No evidence of caries
  * 1 Initial caries
  * 2 Distinct visual change in enamel
  * 3 Localised enamel breakdown due to caries with no visible dentine
  * 4 Underlying dark shadow from dentine
  * 5 Distinct cavity with visible dentine
  * 6 Extensive distinct cavity with visible dentine
Socio-Professional Category | Day 1
  * Farmers,
  * artisans,
  * traders and business leaders,
  * executives and higher intellectual professions,
  * intermediate professions,
  * employees,
  * workers

SECONDARY OUTCOMES:
Communication needed between dentist and orthodontist | At 48 months
  focus group of dentist and orthodontist at the beginning and at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France